CLINICAL TRIAL: NCT01036113
Title: A Phase 2, Open-Label Study of EZN-2208 (PEG-SN38) in Patients With Previously Treated Metastatic Breast Cancer (MBC)
Brief Title: A Phase 2 Study of EZN-2208 in Patients With Metastatic Breast Cancer
Acronym: PEG-SN38
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Program suspended and divested
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EZN-2208-03
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2012-10

CONDITIONS: Metastatic Breast Cancer
Keywords: EZN-2208 (PEG-SN38)
MeSH Terms: conditions — Breast Neoplasms | interventions — EZN-2208

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: EZN-2208 (Experimental): Experimental: EZN-2208 EZN-2208 will be administered as an i.v. infusion on weekly basis for 3 weeks and repeated every 28 days.
  Interventions: Drug: EZN-2208

INTERVENTIONS:
Drug: EZN-2208 — EZN-2208 will be administered as an i.v. infusion on weekly basis for 3 weeks and repeated every 28 days.
  Other Names: Peg SN38

SUMMARY:
This is a Phase 2, multicenter, open-label, noncomparative study to evaluate safety,efficacy and of single-agent EZN 2208 administered in patients with previously treated MBC.

After discontinuation of study treatment, patients will receive care as considered appropriate by the investigator. Patients will continue to be followed for disease progression, subsequent anticancer therapy, and survival.

DETAILED DESCRIPTION:
EZN-2208 will be administered by i.v. infusion weekly for 3 weeks in 4-week cycles. Study treatment will be continued until evidence of disease progression, unacceptable toxicity, or withdrawal of the patient's consent for participation in the study.

Approximately 160 patients with previously treated MBC will be enrolled in this study. Eighty patients in each of two cohorts will be evaluated as follows:

1. AT Cohort - Patients treated with prior anthracycline and taxane as adjuvant or metastatic therapy; no more than 2 prior chemotherapy regimens for MBC
2. ATX Cohort - Patients treated with prior anthracycline, taxane, and Xeloda® (capecitabine) as adjuvant or metastatic therapy; no more than 4 prior chemotherapy regimens for MBC

After discontinuation of study treatment, patients will receive care as considered appropriate by the investigator. Patients will continue to be followed for disease progression, subsequent anticancer therapy, and survival for at least 6 months after enrollment of the last patient in the study

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast adenocarcinoma that is metastatic. Receptor status of the tumor must be known.
* Disease progression during or after immediate previous therapy, or intolerable toxicity leading to cessation of immediate previous therapy
* Previous treatment for MBC:

  * AT Cohort: Prior AT required as adjuvant or metastatic therapy; no more than 2 prior chemotherapy regimens for MBC.
  * ATX Cohort: Prior ATX required as adjuvant or metastatic therapy;no more than 4 prior chemotherapy regimens for MBC.
* For patients with positive receptor status:

  * Patients with HER2+ MBC must have received prior trastuzumab.
  * Patients with ER+ MBC must have received prior hormone therapy.
* Measurable disease by RECIST Version 1.1
* Women 18 years or older
* ECOG performance status of 0 to 2
* Adequate bone marrow, renal and hepatic functions

Exclusion Criteria:

* Major surgery within 3 weeks before study start
* Known or suspected brain metastases requiring intervention with steroids and/or radiation therapy
* Prior chemotherapy, immunotherapy, non-investigational agent, or other therapy used to treat the cancer within 3 weeks before scheduled administration of EZN-2208
* History of other primary cancer within 5 years of enrollment, unless

  1. Curatively resected non-melanomatous skin cancer, or
  2. Curatively resected cervical cancer
* Lack of recovery to Grade 1 from any reversible side effects related to the administration of an investigational agent, chemotherapy, or other prior treatments for the cancer
* Current participation in another clinical study with an investigational agent and/or use of an investigational drug (not including investigational use of an approved drug) in the 30 days before the first administration of EZN-2208
* Known chronic infectious disease, such as AIDS

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Response Rate | 2011

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 2011

CONTACTS AND LOCATIONS:
Overall Officials: Joyce A O'Shaughnessy, MD, Principal Investigator — Texas Oncology-Baylor Charles A. Sarnrnons Cancer Center
Locations (36):
- United States (36):
  - Location #12, Sedona, Arizona
  - Location #5, Tucson, Arizona
  - Location #32, Murrieta, California
  - Location #39, Oxnard, California
  - Location #18, Denver, Colorado
  - Location #36, New Port Richey, Florida
  - Location #1, Ocoee, Florida
  - Location #40, Niles, Illinois
  - Location #15, Carmel, Indiana
  - Location #10, Minneapolis, Minnesota
  - Location #16, Columbia, Missouri
  - Location #14, Kansas City, Missouri
  - Location #2, Henderson, Nevada
  - Location#19, Troy, New York
  - Location #4, Raleigh, North Carolina
  - Location #41, Columbus, Ohio
  - Location #27, Portland, Oregon
  - Location #8, Greenville, South Carolina
  - Location #33, Abilene, Texas
  - Location #34, Arlington, Texas
  - Location #9, Austin, Texas
  - Location #3, Bedford, Texas
  - Location #26, Dallas, Texas
  - Location #13, Dallas, Texas
  - Location #30, Dallas, Texas
  - Location #17, Dallas, Texas
  - Location #24, Fort Worth, Texas
  - Location #11, Houston, Texas
  - Location #38, Lewisville, Texas
  - Location #31, McAllen, Texas
  - Location # 28, Midland, Texas
  - Location #35, Sugar Land, Texas
  - Location# 20, Tyler, Texas
  - Location #23, Fairfax, Virginia
  - Location #7, Norfolk, Virginia
  - Location #21, Salem, Virginia